CLINICAL TRIAL: NCT01586156
Title: Pulmonary Arterial Hypertension Treatment With Carvedilol for Heart Failure
Brief Title: PAHTCH Pulmonary Arterial Hypertension Treatment With Carvedilol for Heart Failure (Carvedilol)
Acronym: PAHTCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Samar Farha, MD, Clinical Study Director, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11-1198; R01HL115008 (NIH)
Record Dates: First submitted 2012-04-23; First posted 2012-04-26 (Estimated); Results first posted 2017-11-30 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-11

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Carvedilol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Open Label Carvedilol (Active Comparator): Eligible subjects will receive open label carvedilol therapy at a dose 3.125 mg twice daily for one week. Subjects will be admitted overnight to the CRU (Clinical Research Unit) for the first-dose challenge of carvedilol. Subjects will take the medication for one week and at the end of one week, eligible subjects will be randomized to one of two groups (blinded). Group 1 will receive 3.125mg twice daily for six months.Group 2 will receive carvedilol in a dose escalation scheme. They will be given 3.125mg tablets to take twice daily for one week, followed by 6.25 mg twice daily for one week, followed by 12.5mg twice daily for one week with the option to increase to the max dose of 25mg twice daily for the remainder of the study.
  Interventions: Drug: Carvedilol
- Placebo Arm (Placebo Comparator): Eligible subjects will receive open label carvedilol therapy at a dose 3.125 mg twice daily for one week. Subjects will be admitted overnight for the first-dose challenge of carvedilol. After one week run in phase, subjects will be placed on placebo. Subjects and Investigators will be blinded to the group assignment for the duration of the study.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Carvedilol — Group 1 will receive 3.125mg carvedilol twice daily for six months.Group 2 will receive carvedilol in a dose escalation scheme.
  Other Names: low fixed dose, escalating dose
  Arms: Open Label Carvedilol
Drug: placebo — Placebo will be taken twice daily for 6 months
  Arms: Placebo Arm

SUMMARY:
Pulmonary arterial hypertension (PAH) is a progressive disease of the pulmonary vasculature leading to elevated pulmonary pressure and right ventricular (RV) dysfunction with heart failure. Measures of RV function are better predictors of mortality and long term outcomes than pulmonary vascular resistance. The interaction between RV function and the pulmonary circulation is not fully understood, but increased after load appears insufficient to explain right heart failure. Yet, all approved PAH therapies target vasodilation of the pulmonary vasculature to lower pressures

DETAILED DESCRIPTION:
Pulmonary arterial hypertension (PAH) is a serious condition characterized by endothelial dysfunction leading to pulmonary vascular constriction, smooth muscle and endothelial proliferation, and progressive right-sided heart failure. The severity of pulmonary hypertension is mostly determined by the response of the right ventricle (RV) to the increased afterload or pulmonary pressures, and RV failure is the leading cause of death in PAH. Most accepted therapies for PAH have been aimed at vasodilation of the pulmonary vasculature, and there has been little thought that PAH patients would benefit from traditional left heart failure treatments. A cornerstone therapy in left heart failure is £]-adrenergic receptor blockade because of its ability to reverse cardiac remodeling and improve clinical outcomes, despite decades of concern regarding its propensity to exacerbate heart failure. It has been reported to reduce mortality by about 30% in patients, and while the precise mechanisms that contribute to its beneficial effects remain to be elucidated, there is evidence that patients with underlying contractile reserve (i.e., via recruitment of viable myocardium with £]-adrenergic receptor stimulation) may experience greater recovery of their cardiac function. In a study using rats with pulmonary hypertension treated with £] blocker, RV function improved, and maladaptive myocardial remodeling was prevented.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 18 or older not greater than age 65 years
* Diagnosis of pulmonary arterial hypertension class 1, 3, 4, 5 (Dana Point 2008)
* NYHA (New York Health Association)/WHO (World Health Organization) Class I-III
* PAH medications must have been initiated according to the latest consensus statement recommendations and remained stable for the last 30 days
* Women of child-bearing age must use a double-barrier local contraception till completion of the study
* Subjects must demonstrate understanding of the study, sign the informed consent, and have a reliable method of communication for contact and ability to comply with the study requirements

Exclusion Criteria:

* Participation in any other treatment studies during enrollment
* Significant illness in the past 30 days requiring hospitalization
* Hepatic insufficiency (transaminase levels > 4 fold the upper limit of normal or bilirubin > 2 fold the upper limit of normal),
* History of HIV, Hepatitis B or C
* Serum creatinine > 2.8 mg/dl
* Pregnancy, breast-feeding, or lack of safe contraception
* Acute decompensated heart failure within past 30 days
* Known allergy or intolerance to carvedilol or other β blockers
* Significant, persistent bradycardia (resting heart rate < 50 bpm) or hypotension (systolic blood pressure < 100 mmHg or mean blood pressure < 70 mmHg) at the time of enrollment
* Second or third-degree AV (Atrial Ventricular) block without pacemaker
* Use of CYP2D6 isoenzyme inhibitors (such as quinidine, fluoxetine, paroxetine, propafenone) which increase drug levels and result in greater vasodilating effects and hypotension
* Use of hypotensive drugs that deplete catecholamines (such as reserpine and monoamine oxidase inhibitors) which may lead to greater signs of hypotension or bradycardia
* Other medical and psychosocial conditions as determined by principal investigator deemed unsuitable for enrollment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-12; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Serpil Erzurum, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

REFERENCES:
- [Result] Farha S, Saygin D, Park MM, Cheong HI, Asosingh K, Comhair SA, Stephens OR, Roach EC, Sharp J, Highland KB, DiFilippo FP, Neumann DR, Tang WHW, Erzurum SC. Pulmonary arterial hypertension treatment with carvedilol for heart failure: a randomized controlled trial. JCI Insight. 2017 Aug 17;2(16):e95240. doi: 10.1172/jci.insight.95240. eCollection 2017 Aug 17. PMID 28814664
- [Result] Saygin D, Highland KB, Farha S, Park M, Sharp J, Roach EC, Tang WHW, Thomas JD, Erzurum SC, Neumann DR, DiFilippo FP. Metabolic and Functional Evaluation of the Heart and Lungs in Pulmonary Hypertension by Gated 2-[18F]-Fluoro-2-deoxy-D-glucose Positron Emission Tomography. Pulm Circ. 2017 Apr-Jun;7(2):428-438. doi: 10.1177/2045893217701917. Epub 2017 Mar 10. PMID 28597761
- [Result] Park JH, Park MM, Farha S, Sharp J, Lundgrin E, Comhair S, Tang WH, Erzurum SC, Thomas JD. Impaired Global Right Ventricular Longitudinal Strain Predicts Long-Term Adverse Outcomes in Patients with Pulmonary Arterial Hypertension. J Cardiovasc Ultrasound. 2015 Jun;23(2):91-9. doi: 10.4250/jcu.2015.23.2.91. Epub 2015 Jun 26. PMID 26140151
- [Derived] Stephens OR, Weiss K, Frimel M, Rose JA, Sun Y, Asosingh K, Farha S, Highland KB, Prasad SVN, Erzurum SC. Interdependence of hypoxia and beta-adrenergic receptor signaling in pulmonary arterial hypertension. Am J Physiol Lung Cell Mol Physiol. 2019 Sep 1;317(3):L369-L380. doi: 10.1152/ajplung.00015.2019. Epub 2019 Jun 26. PMID 31242023
- [Derived] Cheong HI, Farha S, Park MM, Thomas JD, Saygin D, Comhair SAA, Sharp J, Highland KB, Tang WHW, Erzurum SC. Endothelial Phenotype Evoked by Low Dose Carvedilol in Pulmonary Hypertension. Front Cardiovasc Med. 2018 Dec 12;5:180. doi: 10.3389/fcvm.2018.00180. eCollection 2018. PMID 30619887

RESULTS

PARTICIPANT FLOW:
Groups:
- Low-fixed-dose Carvedilol: Eligible subjects will receive open label carvedilol therapy at a dose 3.125 mg twice daily for one week. Subjects will be admitted overnight to the CRU for the first-dose challenge of carvedilol. Subjects will take the medication for one week and at the end of one week, eligible subjects will be randomized to one of two groups (blinded). Group 1 will receive 3.125mg twice daily for six months. This is the low fixed dose Carvedilol
- Placebo Arm: Eligible subjects will receive open label carvedilol therapy at a dose 3.125 mg twice daily for one week. Subjects will be admitted overnight for the first-dose challenge of carvedilol. After one week run in phase, subjects will be placed on placebo. Subjects and Investigators will be blinded to the group assignment for the duration of the study.
  Carvedilol placebo: Placebo taken twice daily for 6 months
- Escalation-dose Carvedilol: Eligible subjects will receive open label carvedilol therapy at a dose 3.125 mg twice daily for one week. Subjects will be admitted overnight to the CRU for the first-dose challenge of carvedilol. Subjects will take the medication for one week and at the end of one week, eligible subjects will be randomized to one of two groups (blinded). Group 2 will receive carvedilol in a dose escalation scheme. They will be given 3.125mg tablets to take twice daily for one week, followed by 6.25 mg twice daily for one week, followed by 12.5mg twice daily for one week with the option to increase to the max dose of 25mg twice daily for the remainder of the study. This is the escalating dose Carvedilol
Period: Overall Study
Arm/Group | Low-fixed-dose Carvedilol | Placebo Arm | Escalation-dose Carvedilol
Started | 10 | 10 | 10
Completed | 10 | 9 | 10
Not Completed | 0 | 1 | 0
Not completed — Pregnancy | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low-fixed-dose Carvedilol | Escalation-dose Carvedilol | Placebo Arm | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 10 | 30
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (6) | 53 (9) | 38 (14) | 42 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 8 | 21
  Male | 3 | 4 | 2 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 10 | 10 | 30
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 4 | 6
  White | 7 | 10 | 6 | 23
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 10 | 10 | 30

OUTCOME MEASURES:

1. Primary Outcome: Cardiac Glucose Uptake in FDG-PET (Fluorodeoxyglucose-Positron Emission Tomography)
Description: We hypothesize that use of carvedilol in patients with PAH (Pulmonary Arterial Hypertension) will decrease the cardiac glucose utilization, and this will be measurable as a drop in fasting FDG-PET standardized uptake values of the heart at 6 months as compared to baseline
Time Frame: 6 months
Population: Paired analyses of baseline to 6 month FDG-PET SUV (standardized uptake value) within each group.
Measure: Median (Inter-Quartile Range); unit: standardized uptake value (SUV)
Arm/Group | Placebo Arm | Low-fixed-dose Carvedilol | Escalation-dose Carvedilol
Number analyzed (Participants) | 10 | 10 | 10
standardized uptake value (SUV)
  baseline FDG-PET | 1.0 [0.6 to 1.4] | 0.6 [0.5 to 0.9] | 0.9 [0.5 to 1.5]
  6 month FDG-PET | 0.8 [0.7 to 1.1] | 0.6 [0.4 to 0.8] | 0.7 [0.4 to 1.0]
Statistical Analysis 1: Comparison: Placebo Arm vs Low-fixed-dose Carvedilol vs Escalation-dose Carvedilol; Test type: Superiority; p = 0.04, ANOVA

2. Secondary Outcome: Urinary cAMP (Cyclic Adenosine Monophosphate)/Creatinine
Description: We hypothesize that use of carvedilol in patients with PAH will increase beta adrenergic receptor function and this will be measurable as an increase in cAMP measured in the urine at 6 months in participants in dose escalation carvedilol.
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: umol/g
Arm/Group | Placebo Arm | Low-fixed-dose Carvedilol | Escalation-dose Carvedilol
Number analyzed (Participants) | 10 | 10 | 10
umol/g
  baseline | 1.4 [1.1 to 1.7] | 0.6 [0.4 to 0.9] | 1.0 [0.6 to 1.1]
  1 month | 1.3 [0.8 to 1.4] | 0.8 [0.5 to 1.1] | 0.7 [0.5 to 0.8]
  3 months | 1.2 [0.8 to 1.8] | 0.6 [0.5 to 1.0] | 1.5 [0.6 to 1.7]
  6 months | 1.4 [0.9 to 2.3] | 0.7 [0.4 to 1.5] | 1.0 [0.8 to 1.4]
Statistical Analysis 1: Comparison: Placebo Arm vs Low-fixed-dose Carvedilol vs Escalation-dose Carvedilol; Test type: Superiority; p = 0.04, ANOVA

3. Secondary Outcome: Beta-Adrenergic Receptor (Alprenolol Binding Assay)
Description: We hypothesize that use of carvedilol in patients with PAH will increase beta- adrenergic receptor availability, and this will be measurable as a increase in alprenolol binding over time of drug use.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: abritrary units
Arm/Group | Placebo Arm | Low-fixed-dose Carvedilol | Escalation-dose Carvedilol
Number analyzed (Participants) | 10 | 10 | 10
abritrary units
  baseline | 92254 (21469) | 85230 (18525) | 82779 (30406)
  6 months | 79083 (22337) | 84554 (22828) | 83730 (20455)
Statistical Analysis 1: Comparison: Placebo Arm vs Low-fixed-dose Carvedilol vs Escalation-dose Carvedilol; Test type: Other — Pearson's correlation test of association of alprenolol binding changes to dose carvedilol; p = 0.02, Pearson — Correlation of the change in alprenolol binding relative to dose carvedilol

4. Other Pre Specified Outcome: Echocardiogram Right Ventricular Systolic Pressure (RVSP)
Description: We hypothesized that RVSP might decrease in participants on carvedilol.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo Arm | Low-fixed-dose Carvedilol | Escalation-dose Carvedilol
Number analyzed (Participants) | 10 | 10 | 10
mm Hg
  baseline | 76 (22) | 63 (28) | 63 (31)
  3 months | 78 (21) | 59 (18) | 54 (24)
  6 months | 66 (23) | 51 (22) | 64 (32)
Statistical Analysis 1: Comparison: Placebo Arm vs Low-fixed-dose Carvedilol vs Escalation-dose Carvedilol; Test type: Superiority; p = 0.05, ANOVA

5. Other Pre Specified Outcome: 6 Minute Walk Test
Description: We hypothesized that carvedilol would not worsen 6 minute walk distance.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Placebo Arm | Low-fixed-dose Carvedilol | Escalation-dose Carvedilol
Number analyzed (Participants) | 10 | 10 | 10
meters
  baseline | 404 (84) | 504 (93) | 438 (158)
  3 months | 412 (84) | 504 (93) | 438 (159)
  6 months | 453 (60) | 486 (90) | 450 (180)

6. Other Pre Specified Outcome: NT-proBNP (N-terminal Pro-B Type Natriuretic Peptide)
Description: We hypothesized that carvedilol would be safe and tolerable and thus that NT-BNP, a measure of heart failure, would not increase in participants on carvedilol.
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Placebo Arm | Low-fixed-dose Carvedilol | Escalation-dose Carvedilol
Number analyzed (Participants) | 10 | 10 | 10
pg/ml
  baseline | 170 [37 to 492] | 57 [28 to 167] | 127 [14 to 518]
  1 month | 183 [68 to 370] | 92 [69 to 208] | 120 [74 to 639]
  3 months | 152 [41 to 487] | 79 [36 to 138] | 169 [50 to 467]
  6 months | 293 [59 to 495] | 52 [32 to 124] | 146 [55 to 348]
Statistical Analysis 1: Comparison: Placebo Arm vs Low-fixed-dose Carvedilol vs Escalation-dose Carvedilol; Test type: Other; p > 0.05, ANOVA

7. Other Pre Specified Outcome: Echocardiogram Left Ventricular Cardiac Output
Description: We hypothesized that carvedilol would be safe and tolerable and thus that Left ventricular cardiac output, a measure of heart function, would not decrease in participants on carvedilol.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Placebo Arm | Low-fixed-dose Carvedilol | Escalation-dose Carvedilol
Number analyzed (Participants) | 10 | 10 | 10
L/min
  baseline | 4.7 (1.7) | 5.2 (2) | 4.5 (0.9)
  3 months | 4.7 (1.2) | 4.6 (1.2) | 4.8 (1.1)
  6 months | 4.5 (0.9) | 4.7 (1.6) | 4.9 (1.7)
Statistical Analysis 1: Comparison: Placebo Arm vs Low-fixed-dose Carvedilol vs Escalation-dose Carvedilol; Test type: Non-Inferiority — Carvedilol did not lead to worse cardiac output as compared to placebo; p = 0.8, ANOVA

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during the duration the subject was consented to participate in the study; 24 weeks or until discontinuation
Description: the definition of adverse event and/or serious adverse event reporting does not differ from the definition listed
Arm/Group | Placebo Arm | Low-fixed-dose Carvedilol | Escalation-dose Carvedilol
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 1/10 | 3/10
Other Adverse Events (participants affected / at risk) | 2/10 | 2/10 | 7/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Arm (N=10) | Low-fixed-dose Carvedilol (N=10) | Escalation-dose Carvedilol (N=10)
Chest pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — Chest pain attributed to pulmonary hypertension
Dyspnea/wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) — Asthma attack brought on from stressor
Leg swelling (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea/vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — complications to chemotherapy
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Arm (N=10) | Low-fixed-dose Carvedilol (N=10) | Escalation-dose Carvedilol (N=10)
Fatigue/vivid dreams (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — shortness of breath due to allergies and weather
Cough/leg swelling (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Blurry vision (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — sinusitis/bronchitis
Broken arm (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — due to fall and unrelated
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Site infection/acute bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Bloating (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) — in association with menstruation
Leg swelling (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
We thought that there would be a possible limitation of hypotension that might limit dosage

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-06-26): https://cdn.clinicaltrials.gov/large-docs/56/NCT01586156/Prot_SAP_000.pdf